CLINICAL TRIAL: NCT05110573
Title: Morbidity and Survival After Minimally Invasive Versus Open Pancreatoduodenectomy: Propensity Score Matched Comparison
Brief Title: Single-centre Propensity Score-matched Comparison of Laparoscopic Versus Open Pancreatoduodenectomy
Acronym: PSMLOPD
Status: Completed | Type: Observational
Sponsor: General Hospital Groeninge (Other)
Responsible Party: Principal Investigator, Dr. M. D'hondt, Dr. Mathieu D'Hondt, Principal investigator, General Hospital Groeninge
Other Study IDs: B3962020000032
Record Dates: First submitted 2021-08-30; First posted 2021-11-08 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-10

CONDITIONS: Pancreatic Neoplasms
Keywords: pancreatoduodenectomy; minimally-invasive surgery; pancreatic cancer; chronic pancreatitis
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatitis, Chronic | interventions — Pancreaticoduodenectomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Laparoscopic pancreatoduodenectomy: Cohort of patients that underwent a Whipple-procedure through a laparoscopic approach.
  Interventions: Procedure: pancreatoduodenectomy
- Open pancreatoduodenectomy: Cohort of patients that underwent a Whipple-procedure through a traditional open approach.
  Interventions: Procedure: pancreatoduodenectomy

INTERVENTIONS:
Procedure: pancreatoduodenectomy — Patients included in the cohorts all underwent pancreatoduodenectomy, open or laparoscopic

SUMMARY:
Minimally invasive pancreatoduodenectomy is increasingly performed. However, technical challenges and a perceived higher risk of complications has hindered wide adoption of a minimally invasive approach.

This is a retrospective comparison of a prospectively kept database. The investigators compared surgical outcomes and survival after laparoscopic (LPD) versus open pancreatoduodenectomy (OPD). In order to reduce the effect of bias and confounding, baseline characteristics of both groups were matched using propensity score matching.

DETAILED DESCRIPTION:
All pancreatoduodenectomies were retrieved from a prospectively kept database and retrospectively analysed. All procedures were performed in a single supra-regional Belgian centre.

The primary endpoint was the major complication rate, defined by a Clavien-Dindo morbidity classification grade IIIa or higher [11]. Secondary endpoints were 90-day mortality rate, length of hospital stay, operative time, blood loss, transfusion requirements and specific pancreatic complications (pancreatic fistula, haemorrhage, and delayed gastric emptying). In addition, overall survival (OS) and disease-free survival (DFS) were analysed in the subgroups of cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of lesion of pancreatic head or peri-ampullary organs

Exclusion Criteria:

* < 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Indications for surgery were benign or malignant lesions of the pancreatic head or peri-ampullary organs. All patients of ≥18 years old diagnosed with suspicious lesions located in the pancreas, ampulla, duodenum or distal bile duct were presented at the multidisciplinary oncological team. In case of biopsy-proven malignancy or clinical and radiological suspicion without confirmed malignancy, surgical resection was considered in accordance with contemporary guidelines
Sampling Method: Non-Probability Sample
Enrollment: 172 (Actual)
Dates: Start 2000-01-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2021-03-20 (Actual)

PRIMARY OUTCOMES:
Major complication rate | 90 days postoperative
  Complications classified as morbidity classification 3a or greater (Clavien-Dindo)

SECONDARY OUTCOMES:
Perioperative outcomes | Up to 30 days
  Operative time (min), blood transfusion requirements, estimated blood loss (mL)
Short-term postoperative outcomes | Up to 30 days
  Hospital stay (days), drain in situ (days), ICU stay (days)
Postoperative morbidity | 90 days
  All complications classified as morbidity classification 3a or greater (Clavien-Dindo)
Pancreatectomy-specific complications | 90 days
  Postoperative pancreatic fistula, Post-pancreatectomy haemorrhage, delayed gastric emptying, as defined by the respective ISGPS classification
Overall survival and disease-free survival | Up to 20 years
  The Kaplan-Meier method was used for estimation of survival and compared between subgroups of cancer patients
Oncological outcomes | Up to 20 years
  Analysis of resection specimen following contemporary pathlogy guidelines and defined by TNM staging system of pancreatic cancer by AJCC/UICC.

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu D'Hondt, MD, Principal Investigator — 1. Department of Digestive and Hepatobiliary/Pancreatic Surgery AZ Groeninge
Locations (1):
- General Hospital Groeninge, Kortrijk, Belgium

REFERENCES:
- [Derived] Vandeputte M, Vansteenkiste F, Ceelen W, De Meyere C, D'Hondt M. Morbidity and survival after laparoscopic versus open pancreatoduodenectomy: propensity score matched comparison. Langenbecks Arch Surg. 2023 Jan 10;408(1):16. doi: 10.1007/s00423-023-02758-y. PMID 36624235